CLINICAL TRIAL: NCT04332679
Title: Guided Bone Regeneration With Non-resorbable Membranes Versus Titanium Meshes and Resorbable Membranes.
Brief Title: Non-resorbable Membranes Versus Titanium Meshes and Resorbable Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GBR Academy (Network)
Responsible Party: Principal Investigator, Alessandro Cucchi, Doctor, GBR Academy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMF 01/2013
Record Dates: First submitted 2020-03-26; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Surgical Procedure, Unspecified; Soft Tissue Infections; Bone Density; Bone Loss; Dental Implant
MeSH Terms: conditions — Soft Tissue Infections; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) The surgeon is masked until the envelope is opened at the time of the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - control group (Active Comparator): 20 patients treated by means of a dense PTFE (d-PTFE) titanium-reinforced membrane (Cytoplast Ti-250XL; Osteogenics Biomedical) and simultaneous implants placement (BT SAFE; Biotec srl, Vicenza, Italy).
  Interventions: Device: Group A - control group
- Group B - Test group (Experimental): 20 patients treated by means of Ti mesh (Trinon Titanium; Karlsruhe, Germany) and cross-linked collagen membrane (Osseoguard, Zimmer Biomet, Warsaw, IN, USA) and simultaneous implants placement (BT SAFE; Biotec srl, Vicenza, Italy).
  Interventions: Device: Group B - Test group

INTERVENTIONS:
Device: Group A - control group — 20 patients treated by means of a dense PTFE (d-PTFE) titanium-reinforced membrane (Cytoplast Ti-250XL; Osteogenics Biomedical) and simultaneous implants placement (BT SAFE; Biotec srl, Vicenza, Italy).
  Arms: Group A - control group
Device: Group B - Test group — 20 patients treated by means of Ti mesh (Trinon Titanium; Karlsruhe, Germany) and cross-linked collagen membrane (Osseoguard, Zimmer Biomet, Warsaw, IN, USA) and simultaneous implants placement (BT SAFE; Biotec srl, Vicenza, Italy).
  Arms: Group B - Test group

SUMMARY:
The objective of this study is to compare two surgical techniques for the treatment of the mandibular bone atrophies: Dense PTFE titanium-reinforced membranes (Group A) versus Titanium mesh covered with cross-linked collagen membranes (Group B).

Therefore, the main purposes are to compare test and control regarding (i) the percentage of post-operative complications (ii) the three-dimensional bone gain (iii) histological, histomorphometrical and microCT outcomes (iv) perImplant bone loss and soft tissue parameters.

DETAILED DESCRIPTION:
In the last 10 years, short- and long-term studies have demonstrated that GBR is a successful and reliable technique for vertical and horizontal ridge augmentation. GBR can be achieved with two different approaches: application of either a polytetrafluoroethylene (PTFE) titanium-reinforced membrane (i.e., a non-resorbable membrane) or a collagen membrane (i.e., a resorbable membrane). To achieve vertical bone augmentation, a resorbable membrane must be supported by a space-making device, such as a titanium mesh (Ti mesh) or a titanium osteosynthesis plate.

However, the use of a barrier device is a technique-sensitive procedure that is not free of complications. The main cause of GBR failure is related to early or late exposure of a barrier device, leading to contamination and infection of the biomaterial, irreversibly compromising bone regeneration.

This study aims to evaluate complication rates and vertical bone gain (VBG) after GBR with dense PTFE titanium-reinforced membranes versus with titanium mesh covered with cross-linked collagen membranes.

The primary objective of the study is, therefore, the evaluation of the healing complications; in particular, the early or delayed exposure of medical devices used for bone regeneration, during the healing period. This exposure is, as reported in all clinical studies, the main cause of the failure of the surgery. A secondary objective, is the quantitative assessment of bone regeneration obtained by the 2 techniques. In particular, the evaluation of the reconstructed bone volume (RBV) with respect to the planned bone volume (PBV). Other targets include the qualitative evaluation of bone regeneration through histological and histomorphometric analysis of the bone biopsies obtained at the moment that the medical device is removed and finally the evaluation of the peri-implant bone resorption will be conducted over time. This study was designed as a pilot, parallel-group, double-blind, randomized, comparative clinical trial. The study was conducted in accordance with the principles of the Declaration of Helsinki. The study was approved by the Ethical Committee of the Sant'Orsola-Malpighi Hospital (Prot. CMF 01/2013; number 30/2013/O/Disp).

The study included 40 patients with partial edentulism, associated with alveolar atrophy in the posterior regions of the mandible, who were referred to the Unit of Oral and Maxillofacial Surgery, Alma Mater Studiorum, University of Bologna, Italy.

Patients were randomized into two study groups, depending on a previous computer-generated randomization sequence. Group A included 20 patients treated by means of a dense PTFE (d-PTFE) titanium-reinforced membrane, and Group B included 20 patients treated by means of a titanium mesh (Ti mesh) and cross-linked collagen membrane.

The study included 3 different treatment phases: the first phase (T0) involves bone regeneration with Dense PTFE titanium-reinforced membranes (Group A) or Titanium mesh covered with cross-linked collagen membranes (Group B) and simultaneous implants placement; the second one (T1), subsequently, after 6 months, this will forsee the removal of the regeneration devices; the third (T2), 3 months after the aforementioned, will forsee the final functional loading of the implants, with a consequent follow-up of the regenerated bone. All the materials and tools used in the study are CE certified and have already been used in the normal care path for patients who have undergone bone regeneration. Moreover, the control visits and the radiological investigations of the data were summarized in the case report form (CRF), and are those that characterize the normal care path of patients undergoing necessary bone regeneration for prosthetic implant rehabilitation when the bone quantity is insufficient.

The primary objective of this study is to evaluate the non-inferiority of group B (Ti mesh) compared to technique A (d-PTFE membrane) in the incidence of complications. The Secondary objectives include: assessment of reconstructed bone volume (RBV) compared to planned bone volume (PBV), histological and histomorphometric analysis of bone quality obtained and periimplant bone resorption after 12 months of follow-up.

The sample size calculation showed that with a minimum of 17 patients per group (total of 34 patients), it will be possible to detect a 35% difference in complications and a difference of 1 mm in VBG between the two groups with a standard deviation a=1 and a significance level of a = 0.05 with a power of 80%. To protect from possible drop-outs, the sample size was increased by to 20 patients per group (total of 40 patients).

The results obtained in the two study groups (Groups A and B) were subjected to statistical description and analyses using specific tests to determine statistically significant differences between them. Both the intent-to-treat and per-protocol populations were analyzed. The patient was regarded as the statistical unit of analysis for all analyses, except that of implant stability, which was carried out considering the implant as the statistical unit. Statistical differences in complication rates were investigated using Fisher's exact test. Differences in implant stability, peri-implant bone defects, and VBG at T0 and T1 were investigated using t-tests for unpaired data. Statistical significance was set at α = 0.05. The statistician was blinded and external to working group.

ELIGIBILITY:
Inclusion Criteria:

* edentulism in posterior regions of the mandible with vertical and horizontal bone resorption of the alveolar ridge requiring three-dimensional bone regeneration and implant-supported rehabilitation
* a vertical peri-implant bone defect of ≥ 2 mm in the alveolar ridge that must be regenerated after placement of implants in a three-dimensional 'ideal' position;
* capacity to understand and accept the conditions of the study; and 4 continuing participation in the study for at least 1 year of follow up.

Exclusion Criteria:

* residual bone height < 5 mm;
* insufficient oral hygiene;
* a smoking habit of > 10 cigarettes/day;
* abuse of alcohol or drugs;
* pregnancy;
* acute local or systemic infection;
* uncontrolled diabetes or other metabolic disease;
* severe hepatic or renal dysfunction; HIV, HBV, or HCV;
* chemotherapy or radiotherapy within the last 5 years;
* immunosuppression therapy;
* autoimmune disorders;
* bisphosphonate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The rate of healing complications after reconstructive surgery | 6 months
  Healing complications are evaluated based on the chronological order in which they occur:• immediate exposure occurs within the 1st month
  * early exposure occurs between the 1st and the 3rd month
  * late exposure occurs between after the 3rd month Evaluation of low-grade and high-grade infection of medical devices used for bone regeneration.
  The former complications are classified as:
  * Class A, including flap damage (soft tissue perforation or laceration)
  * Class B, including neurological damage (paresthesia or disesthesia)
  * Class C,including vascular damage (hemorrhage). The latter complications are divided into four classes, according to the presence and extent of exposure, as well as the presence of a purulent exudate:
  * Class I, membrane exposure <3 mm, no purulent exudate
  * Class II membrane exposure >=3mm, no purulent exudate
  * Class III: membrane exposure, with purulent exudate

SECONDARY OUTCOMES:
Implants Insertion Torque | during surgery
  measured with a manual dynamometric torque wrench, able to measure torques up to 100 Ncm
Change in implant Stability | during surgery/after 6 months
  Change from implant stability during surgery and at 6 months was evaluated using the implant stability quotient recorded during surgery and after 6 months during reopening surgery
Vertical bone gain | at 6 months
  calculated as the difference between the initial bone defect and the residual bone defect expressed in millimeters (mm).
Bone tissue area (B.ar) | at 6 months
  evaluated as the total area of regenerated bone performed with a digital microscopic evaluation.
Bone volume (B.V) | at 6 months
  evaluated as the total volume of the regenerated bone performed with a MicroCT evaluation.
Peri-implant bone level (PBL) | at 1 years
  was evaluated as the distance between the implant shoulder and the visible bone crest on periapical radiograph using a parallel technique. The distance was measured to the nearest 0.01 mm using an image analysis software (Image J, NIH).
Inter-proximal bone peaks (IBP) | at 1 years
  was evaluated as the distance between the interproximal bone peak and the "ideal" regeneration line on periapical radiograph using a parallel technique. The distance was measured to the nearest 0.01 mm using an image analysis software (Image J, NIH)
Probing pocket depth (PPD) | at 1 years
  The probing depth was measured from the gingival margin at the base of the groove or pocket in the central and distal mesial sites, using the calibrated Click-probe millimeter probe 3/5/7/10 mm scale
Thickness of keratinized tissue (tKT) | at 1 years
  The thickness of the soft tissues was determined apically at the gingival margin using a file for endodontic therapy measures 8 and with a 3 mm diameter silicone disk with a stop function
Width of keratinized mucosa (wKT) | at 1 years
  The height of the keratinized mucosa was determined by the gingival margin at the vestibular muco-gingival line

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Corinaldesi, Study Director — unibo
Locations (1):
- School of Dentistry - University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Original articles in international journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: june 2020
Access Criteria: Access credentials to journal resources

REFERENCES:
- [Derived] Cucchi A, Vignudelli E, Fiorino A, Pellegrino G, Corinaldesi G. Vertical ridge augmentation (VRA) with Ti-reinforced d-PTFE membranes or Ti meshes and collagen membranes: 1-year results of a randomized clinical trial. Clin Oral Implants Res. 2021 Jan;32(1):1-14. doi: 10.1111/clr.13673. Epub 2020 Oct 19. PMID 33017060